CLINICAL TRIAL: NCT04463134
Title: A Prospective Observational Study of Parameters Related to the Clinical Outcomes of NTM Pulmonary Disease in Prince of Wales Hospital
Brief Title: An Observational Study on Patients With NTM Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, LAI PING LO, Resident, Chinese University of Hong Kong
Other Study IDs: 2020.123
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Clinical Outcomes
Keywords: Disease progression, death
MeSH Terms: conditions — Disease Progression; Death | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: They will start pharmacological treatment according to guidelines and sensitivity
  Interventions: Drug: NTM drug treatment
- Observation group: They will not start pharmacological treatment. They will be monitored on symptoms, sputum conversion and radiological progression

INTERVENTIONS:
Drug: NTM drug treatment — NTM drug treatment according to guideline and sensitivity test results
  Other Names: pharmacological treatment
  Groups: Treatment group

SUMMARY:
Non-tuberculous mycobacterial (NTM) infection is becoming more and more common, especially causing pulmonary diseases in those elderly or the immunocompromised. The diagnosis, treatment and monitoring of NTM pulmonary disease(NTMPD) are not updated and real life management if also challenging.

DETAILED DESCRIPTION:
Non-tuberculous mycobacteria (NTM) are a large group of ubiquitous microorganisms in the natural environment as well as household water systems . Over 180 different species have been identified but only 32 are reported to cause diseases in human or animals. NTM infection can affect the lung, skin and soft tissue, lymph node or cause disseminated diseases in the immunocompromised. NTM pulmonary diseases are the most important disease entity, accounting for 75-94% of all clinically important NTM cases.

The predominant species and their pathogenicity vary in different countries. While Mycobacterium avium-intracellulare complex (MAC) is most prevalent in the USA, Canada, Australia, Japan, Taiwan and Hong Kong, M. abscessus complex is more common in Singapore and M. Kansasii in European counties, respectively. Recently reports showed an increasing trend in importance of NTM PD in a few countries.

NTM can cause chronic and debilitating pulmonary disease with increased morbidity and even mortality. Healthy individuals can be affected though many have underlying structural lung diseases or immunodeficient conditions. Patients usually present with nonspecific symptoms, including productive cough, dyspnea, hemoptysis, fever, weight loss and malaise. Therefore, the diagnosis of NTM pulmonary disease (NTMPD) is challenging requiring comprehensive clinical, microbiological and radiological data according to in the American Thoracic Society and Infectious Diseases Society of America (ATS/IDSA) 2007 guidelines. Treatment of NTMPD is also a difficult decision because some remain stable for a long period without treatment while the others progress to severe and even fatal diseases. A prolonged course of antibiotic involving multiple agents with potential adverse effects is needed but a cure cannot be guaranteed. Moreover, the treatment regimens might be different from those recommended by the international guidelines after balancing multiple factors, including patients' comorbidities, disease severity, and the species and antimicrobial susceptibility of the causative organism. Therefore, whom to treat, when to start and how to treat is a clinical dilemma. Epidemiological data of NTM remains unclear although an increase in prevalence and incidence are consistently observed globally. It is not a notifiable disease in most of the countries and data mainly comes from sentinel surveillance and microbiological results.

Local epidemiological data of NTM infection in Hong Kong is largely scarce apart from a small study done 25 years ago in 1995. Further local investigation on the epidemiology, disease course and clinical practice is needed to optimize their management.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or above
* Two or more respiratory samples positive for NTM, including sputum, tracheal aspirates, bronchial washing, bronchial aspirates, bronchial trap and bronchoalveolar lavage or lung biopsy

Exclusion Criteria:

* NTM isolates from extrapulmonary samples
* Refused to sign an informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suspected NTMPD followed up in the Prince of Wales Hospital will be recruited
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes of NTMPD patients with or without treatment in 1 year | 1 year
  Clinical outcomes include stable disease, disease progression, chest infection, death.

SECONDARY OUTCOMES:
Clinical parameters that predict the disease progression | 1 year
  Clinical parameters include demographics and comorbidities.
Functional | 1 year
  functional capacity of patients including mobility, exercise tolerance, lung function
Microbiological parameters that predict disease progression | 1 year
  species subtypes, smear positivity and drug resistance
Radiological features that predict disease progression | 1 year
  Pattern and extent of lung involvement

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Falkinham JO 3rd. Environmental sources of nontuberculous mycobacteria. Clin Chest Med. 2015 Mar;36(1):35-41. doi: 10.1016/j.ccm.2014.10.003. Epub 2014 Nov 6. PMID 25676517
- [Background] Gebert MJ, Delgado-Baquerizo M, Oliverio AM, Webster TM, Nichols LM, Honda JR, Chan ED, Adjemian J, Dunn RR, Fierer N. Ecological Analyses of Mycobacteria in Showerhead Biofilms and Their Relevance to Human Health. mBio. 2018 Oct 30;9(5):e01614-18. doi: 10.1128/mBio.01614-18. PMID 30377276
- [Background] Gupta RS, Lo B, Son J. Phylogenomics and Comparative Genomic Studies Robustly Support Division of the Genus Mycobacterium into an Emended Genus Mycobacterium and Four Novel Genera. Front Microbiol. 2018 Feb 13;9:67. doi: 10.3389/fmicb.2018.00067. eCollection 2018. PMID 29497402
- [Background] Henkle E, Winthrop KL. Nontuberculous mycobacteria infections in immunosuppressed hosts. Clin Chest Med. 2015 Mar;36(1):91-9. doi: 10.1016/j.ccm.2014.11.002. Epub 2014 Dec 23. PMID 25676522
- [Background] Johnson MM, Odell JA. Nontuberculous mycobacterial pulmonary infections. J Thorac Dis. 2014 Mar;6(3):210-20. doi: 10.3978/j.issn.2072-1439.2013.12.24. PMID 24624285
- [Background] Zweijpfenning SMH, Ingen JV, Hoefsloot W. Geographic Distribution of Nontuberculous Mycobacteria Isolated from Clinical Specimens: A Systematic Review. Semin Respir Crit Care Med. 2018 Jun;39(3):336-342. doi: 10.1055/s-0038-1660864. Epub 2018 Aug 2. PMID 30071548
- [Background] Prevots DR, Shaw PA, Strickland D, Jackson LA, Raebel MA, Blosky MA, Montes de Oca R, Shea YR, Seitz AE, Holland SM, Olivier KN. Nontuberculous mycobacterial lung disease prevalence at four integrated health care delivery systems. Am J Respir Crit Care Med. 2010 Oct 1;182(7):970-6. doi: 10.1164/rccm.201002-0310OC. Epub 2010 Jun 10. PMID 20538958
- [Background] Namkoong H, Kurashima A, Morimoto K, Hoshino Y, Hasegawa N, Ato M, Mitarai S. Epidemiology of Pulmonary Nontuberculous Mycobacterial Disease, Japan. Emerg Infect Dis. 2016 Jun;22(6):1116-7. doi: 10.3201/eid2206.151086. No abstract available. PMID 27191735
- [Background] Kim HO, Lee K, Choi HK, Ha S, Lee SM, Seo GH. Incidence, comorbidities, and treatment patterns of nontuberculous mycobacterial infection in South Korea. Medicine (Baltimore). 2019 Nov;98(45):e17869. doi: 10.1097/MD.0000000000017869. PMID 31702652
- [Background] Morimoto K, Iwai K, Uchimura K, Okumura M, Yoshiyama T, Yoshimori K, Ogata H, Kurashima A, Gemma A, Kudoh S. A steady increase in nontuberculous mycobacteriosis mortality and estimated prevalence in Japan. Ann Am Thorac Soc. 2014 Jan;11(1):1-8. doi: 10.1513/AnnalsATS.201303-067OC. PMID 24102151
- [Background] Vinnard C, Longworth S, Mezochow A, Patrawalla A, Kreiswirth BN, Hamilton K. Deaths Related to Nontuberculous Mycobacterial Infections in the United States, 1999-2014. Ann Am Thorac Soc. 2016 Nov;13(11):1951-1955. doi: 10.1513/AnnalsATS.201606-474BC. PMID 27607541
- [Background] Griffith DE, Aksamit T, Brown-Elliott BA, Catanzaro A, Daley C, Gordin F, Holland SM, Horsburgh R, Huitt G, Iademarco MF, Iseman M, Olivier K, Ruoss S, von Reyn CF, Wallace RJ Jr, Winthrop K; ATS Mycobacterial Diseases Subcommittee; American Thoracic Society; Infectious Disease Society of America. An official ATS/IDSA statement: diagnosis, treatment, and prevention of nontuberculous mycobacterial diseases. Am J Respir Crit Care Med. 2007 Feb 15;175(4):367-416. doi: 10.1164/rccm.200604-571ST. No abstract available. PMID 17277290
- [Background] Hwang JA, Kim S, Jo KW, Shim TS. Natural history of Mycobacterium avium complex lung disease in untreated patients with stable course. Eur Respir J. 2017 Mar 8;49(3):1600537. doi: 10.1183/13993003.00537-2016. Print 2017 Mar. PMID 28275170
- [Background] Park J, Cho J, Lee CH, Han SK, Yim JJ. Progression and Treatment Outcomes of Lung Disease Caused by Mycobacterium abscessus and Mycobacterium massiliense. Clin Infect Dis. 2017 Feb 1;64(3):301-308. doi: 10.1093/cid/ciw723. Epub 2016 Nov 10. PMID 28011609
- [Background] Igari H, Yamagishi K, Yamazaki S, Murata S, Yahaba M, Takayanagi S, Kawasaki Y, Taniguchi T. A retrospective observational study of antimicrobial treatment for non-tuberculous mycobacteria disease using a nationwide claims database in Japan. J Infect Chemother. 2020 Apr;26(4):349-352. doi: 10.1016/j.jiac.2019.10.009. Epub 2019 Nov 11. PMID 31727566
- [Background] van Ingen J, Wagner D, Gallagher J, Morimoto K, Lange C, Haworth CS, Floto RA, Adjemian J, Prevots DR, Griffith DE; NTM-NET. Poor adherence to management guidelines in nontuberculous mycobacterial pulmonary diseases. Eur Respir J. 2017 Feb 15;49(2):1601855. doi: 10.1183/13993003.01855-2016. Print 2017 Feb. No abstract available. PMID 28182571
- [Background] Adjemian J, Olivier KN, Seitz AE, Holland SM, Prevots DR. Prevalence of nontuberculous mycobacterial lung disease in U.S. Medicare beneficiaries. Am J Respir Crit Care Med. 2012 Apr 15;185(8):881-6. doi: 10.1164/rccm.201111-2016OC. Epub 2012 Feb 3. PMID 22312016
- [Background] Shah NM, Davidson JA, Anderson LF, Lalor MK, Kim J, Thomas HL, Lipman M, Abubakar I. Pulmonary Mycobacterium avium-intracellulare is the main driver of the rise in non-tuberculous mycobacteria incidence in England, Wales and Northern Ireland, 2007-2012. BMC Infect Dis. 2016 May 6;16:195. doi: 10.1186/s12879-016-1521-3. PMID 27154015
- [Background] Thomson R, Donnan E, Konstantinos A. Notification of Nontuberculous Mycobacteria: An Australian Perspective. Ann Am Thorac Soc. 2017 Mar;14(3):318-323. doi: 10.1513/AnnalsATS.201612-994OI. PMID 28118021
- [Background] Ide S, Nakamura S, Yamamoto Y, Kohno Y, Fukuda Y, Ikeda H, Sasaki E, Yanagihara K, Higashiyama Y, Hashiguchi K, Futsuki Y, Inoue Y, Fukushima K, Suyama N, Kohno S. Epidemiology and clinical features of pulmonary nontuberculous mycobacteriosis in Nagasaki, Japan. PLoS One. 2015 May 28;10(5):e0128304. doi: 10.1371/journal.pone.0128304. eCollection 2015. PMID 26020948
- [Background] Ding LW, Lai CC, Lee LN, Hsueh PR. Disease caused by non-tuberculous mycobacteria in a university hospital in Taiwan, 1997-2003. Epidemiol Infect. 2006 Oct;134(5):1060-7. doi: 10.1017/S0950268805005698. Epub 2006 Feb 22. PMID 16492317
- [Background] Park YS, Lee CH, Lee SM, Yang SC, Yoo CG, Kim YW, Han SK, Shim YS, Yim JJ. Rapid increase of non-tuberculous mycobacterial lung diseases at a tertiary referral hospital in South Korea. Int J Tuberc Lung Dis. 2010 Aug;14(8):1069-71. PMID 20626955
- [Background] Stout JE, Koh WJ, Yew WW. Update on pulmonary disease due to non-tuberculous mycobacteria. Int J Infect Dis. 2016 Apr;45:123-34. doi: 10.1016/j.ijid.2016.03.006. Epub 2016 Mar 11. PMID 26976549